CLINICAL TRIAL: NCT04483752
Title: Predicting the Progression to Chronic Fibrosis of Lung Lesions Related to Covid-19 Infection From Chest CT Images
Acronym: PREDISCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A01322-37
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: CoV2 SARS Pneumonia
Keywords: SARS CoV2; COVID-19; fibrosis
MeSH Terms: conditions — COVID-19; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalised for SARS CoV-2 infection. (Other)
  Interventions: Other: CHEST CT SCAN

INTERVENTIONS:
Other: CHEST CT SCAN — Chest CTscan at 3 and 12 months

SUMMARY:
The main differences observed between SARSCoV-2 pneumonia and other epidemic viral pneumopathies (e.g., seasonal influenza) are the greater infectivity of SARSCoV-2, the clinical severity of the disease, particularly in young patients without co-morbidities, and the observation of radiological images related to significant parenchymal aggression in a large number of patients.

The lesions in the acute phase correspond essentially to bilateral ground glass opacity more or less associated with condensations which would be markers of more severe infections.

The major scope of the lesions in the acute phase raises the question of whether or not the scanning anomalies are completely resolved over time, and the possible impact on lung function. This risk of sequelae is very important to study given the large number of patients affected by SARSCoV-2, especially since these are often young patients who appear to be "healthy".

In the current context of the CoV-2 SARS pandemic, the improved quality and availability of diagnostic scanners provides a wealth of information on the semiology and progression of lung disease with minimal exposure to ionizing radiation. A majority of hospitalized patients with SARSCoV-2 received a CT scan in the early phase of the disease. Indeed, the French Society of Radiology has recommended the performance of a CT scan without injection in thin sections in case of suspicion or for confirmation of the diagnosis in patients presenting initial or secondary clinical signs of severity and justifying hospital management due to the initial lack of reagents for performing biological tests (RT-PCR) and the high sensitivity of the CT scan and its specificity in epidemic periods.

The present study aims to study the kinetics of lung involvement in SARS CoV 2, to study the predictive character of the chest CT scan performed at the patient's discharge on the existence of radiological sequelae at 3 months but also at 1 year in order not to misunderstand the constitution of late fibrosis after partial resolution of the CT images. The investigatos will study the correlation between possible radiological abnormalities and the clinical presentation (patient symptoms and lung function). The rigorous follow-up of these patients will allow us to set up, if necessary, early treatment of the detected abnormalities (inhaled corticoids in case of bronchial or bronchiolar damage, study of the place of an anti-fibrosis treatment in case of fibrosis,...).

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for SARS CoV-2 infection proved by RT-PCR and/or by a typical SARS CoV-2 pneumonia clinic and imaging that required hospitalization Scan performed when the patient is no longer oxygenating, i.e. at least 48 hours prior to hospital discharge (discharge criterion) up to a maximum of 1 month after hospitalisation.
* Patient ≥ 18 years old
* Patient who has given free, informed and written consent

Exclusion Criteria:

* Patient ≤ 18 years old
* CT Contraindication
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-24 (Estimated); Study Completion 2022-12-24 (Estimated)

PRIMARY OUTCOMES:
description of the different types of lesions | 3 months

SECONDARY OUTCOMES:
quantification of circulating antibodies and correlation between the level of immunization against SARS CoV2, the severity of the initial disease and the existence or not of long-term pulmonary sequelae | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Saint Joseph, Paris
  - Institut Gustave Roussy (IGR), Villejuif